CLINICAL TRIAL: NCT03008720
Title: EVALUATION OF ELECTRICAL ACTIVITY TIBIAL MUSCLE AND POSTURAL CONTROL OF INDIVIDUALS WITH HEMIPARESIA FROM AVE SUBMITTED TDCS ASSOCIATED WITH FES - CLINICAL STUDY, RANDOMIZED, DOUBLE BLIND.
Brief Title: Evaluation of Electrical Activity Tibial Muscle and Postural Control of Individuals With Hemiparesia Post TDCS Associated With FES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Aline Marina Alves Fruhauf, Professor of graduation., University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 767.866
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Hemiparesis; Transcranial Direct Current Stimulation; Electromyography
Keywords: functional electrical simulation
MeSH Terms: conditions — Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- tDCS active (Active Comparator): Transcranial stimulation ( tDCS ) active will be administered using Tct Research 1 CH tdcs Simulator model 101. tDCS will be performed for 20 minutes and intensity 2mA associated active contraction of the TA muscle.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- tDCS sham (Placebo Comparator): Placebo tDCS will follow the same procedures as active tDCS with active, but the tDCS device will only be switched on for 20 seconds.
  Interventions: Device: Sham stimulation
- FES active (Active Comparator): Functional electrical stimulation (FES) active will be administered using QUARK® FES VIF 995 DUAL device. The duration of active FES will be 20 minutes, associated with active contraction of the TA muscle. The pulse width will be 250 μs, modulated at a frequency of 50 Hz, with one to two stimulation cycles (6 seconds on and 12 seconds off) and the intensity will be increased until reaching the motor threshold.
  Interventions: Device: Functional electrical stimulation (FES)
- FES sham (Placebo Comparator): Placebo FES will follow the same procedures as active FES , but the FES device will only be switched on for 20 seconds, following which the intensity will be gradually reduced to 0 mA.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS)
  Arms: tDCS active
Device: Functional electrical stimulation (FES)
  Arms: FES active
Device: Sham stimulation
  Arms: FES sham; tDCS sham

SUMMARY:
Introduction: It is suggested that increased cortical activity, induced by cerebral stimulation associated or not with other rehabilitation techniques, may potentiate the motor and functional therapeutic effects in individuals with neurological deficits. Objectives: To evaluate the electrical activity of the anterior tibial muscle (TA) and postural control of individuals with hemiparesis due to stroke following treatment with transcranial direct current (tDCS) stimulation and functional electrical stimulation (FES), associated or isolated). (EMG) and postural control by the Balance Evaluation Systems Test (BESTest). Both of which were collected at four different time points: pre-treatment, immediately after 10 treatment sessions, and 30 days follow-up after the interventions. Patients will be randomized into 4 experimental groups: tDCS anodic active + active FES+ active contraction TA, tDCS sham + active FES+ active contraction TA, tDCS anodic active+ placebo FES+ active contraction TA, tDCS sham+ FES sham+ active contraction TA. tDCS (2mA) will be applied over the motor (Cz) and cathodic vertex over the supraorbital region of the normal hemisphere and FES over hemiparetic TA by a researcher who will not be the one who will evaluate the anesthesia patient. The treatment will last 10 sessions, twice a week, with a time of 20 minutes.

ELIGIBILITY:
Inclusion criteria:

* Individuals with hemiparesis due to stroke;
* Both sexes;
* Agree to sign the free and informed consent form.

Exclusion criteria:

* Positive cut-off point for the Mini Mental State Examination (MMSE) of less than 11 points already corrected for schooling;
* Ankle mobility reduced by history of fracture or use of ankle fasteners;
* Irreducible equine deformity;
* Muscle strength level of AT less than 1 by the scale of Kendall;
* Patients with reported severe visual impairment;
* Contraindications to the use of transcranial direct current stimulation (history of seizure or recurrent epilepsy, brain tumors at the stimulation site, metallic materials implanted in the brain);
* Individuals with cutaneous infection at the point of application of FECC or FES;
* Individuals who presented anesthesia or hyperesthesia at the point of application of the ECTS;
* Individuals diagnosed with deep venous thrombosis (DVT);
* Individuals diagnosed with degenerative diseases or polyneuropathies.
* Individuals who do not present complementary tests that diagnose the lesion site.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
electrical activity (median frequency and amplitude of the electromyographic signal) of the anterior tibial muscle | 1 YEAR